CLINICAL TRIAL: NCT05151328
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of Plecanatide in the Treatment of Functional Constipation in Chinese Patients for up to 12 Weeks
Brief Title: Efficacy and Safety of Plecanatide Comparing With Placebo in the Treatment of Functional Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Luoxin Pharmaceutical Group Stock Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NC011901
Record Dates: First submitted 2021-11-04; First posted 2021-12-09 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Functional Constipation
MeSH Terms: interventions — plecanatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plecanatide group(n=320) (Experimental): The investigational products are administrated orally, each patient will take one table (Plecanatide 3.0mg) Once daily(QD) in the day before 18:00 with approximately of water. If the investigational product is not taken in the day before 18:00 then skip the dose on that day and take the next dose on the next regular time. The duration of treatment is 12 weeks.
  Interventions: Drug: Plecanatide
- Placebo group (n=320) (Placebo Comparator): The investigational products are administrated orally, each patient will take one table (Placebo 3mg) QD in the day before 18:00 with approximately of water. If the investigational product is not taken in the day before 18:00 then skip the dose on that day and take the next dose on the next regular time. The duration of treatment is 12 weeks.
  Interventions: Drug: Plecanatide

INTERVENTIONS:
Drug: Plecanatide — Plecanatide or Placebo; Route of Plecanatide/placebo administration: tablet; dosage: 3mg, dosage form oral; Frequency of administration: QD
  Other Names: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, Placebo-controlled Phase III clinical study to evaluate the efficacy and safety of Plecanatide in the treatment of Functional Constipation in Chinese patients for up to 12 weeks.

Patients will enter a Screening period which must undergo a 2-week Pre-Treatment assessment, they will complete daily assessments of electronic dairy to demonstrate the eligibility.

Eligible subjects will be randomized into Plecanatide 3 mg group or Placebo group at Visit 1 at the ratio of 1:1 and take an oral dose of study treatment continuously for 12 weeks. For 2 weeks after complete dosing patients will continue to complete daily electronic dairy. Patients will then return to the clinical site for efficacy and safety assessment as part of an End of Study visit. The planned duration of participation in this study will be 154 days and up to 164 days with all windows considered.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing and able to participate in the study for the required duration, can understand and is willing to sign the （Inform Consent Form)ICF and agrees to undergo all protocol-related tests and procedures.
2. Males or females over 18 years of age (inclusive) when signed the （Inform Consent Form)ICF.
3. Patient agrees to use adequate medical contraception from signing of informed consent through 28 days after the first dose of study drug
4. Colonoscopy with normal or mildly abnormal results.
5. Patient meets the Rome Ⅳ functional constipation criteria as modified for this study for at least 3 months prior to the Screening visit with symptom onset for at least 6 months prior to the diagnosis. The Rome Ⅳ criteria as modified for this study require the following:
6. Patients who meet the modified Rome Ⅳ criteria based on history must also demonstrate the following during the two-week Pre-Treatment Electronic hand-held device(EHD) assessment period.
7. Patient must complete at least 6 of the 7 daily (Electronic Diary) eDiary entries during each week of the 2-week pre-treatment assessment period.
8. Patient is able to communicate with Investigator and understand and comply with scheduled visits, study treatment, laboratory tests, and other study-related procedures and requirements during the study.

Exclusion Criteria:

1. Previous use of Plecanatide.
2. Previous anaphylactic reaction to any medication.
3. Females are excluded if lactating.
4. Patient has unexplained and clinically significant "alarm symptoms" including nonhemorrhoidal lower Gastrointestinal (GI) bleeding, iron-deficiency anemia, weight loss.
5. Patient with known constipation due to secondary causes.
6. Patient had a known structural abnormality of the gastrointestinal tract or a condition that may affect gastrointestinal motility or defecation
7. Patient had a history of chronic disease with abdominal pain or discomfort that would interfere with the evaluation of this study
8. Patient has active peptic ulcer.
9. Patient has had or is scheduled to have abdominal surgery during the study.
10. Patient has fecal impaction requiring hospitalization or emergency room treatment.
11. Patient has traveled to a region considered as high risk for developing traveler's diarrhea while participating in the study.
12. Patient has a history of cancer (other than basal cell or squamous cell carcinoma of the skin) unless the malignancy has been in a complete remission without maintenance chemotherapy for at least 5 years prior to the Screening visit.
13. Known or suspected alcoholism or drug addiction or significant drug abuse within 1 year of the Screening visit.
14. Patient has a history of diabetic neuropathy.
15. Patient has hypothyroidism.
16. Patient has active HBV、HCV or HIV antibody positive.
17. Patient with severe cardiopulmonary or other organ dysfunction.
18. Patient with significant abnormalities in physical examination, ECG, or laboratory tests that, in the judgment of the investigator, would make the patient inappropriate for this study.
19. Evaluation of BSFS not met before administration。
20. Patient uses Dulcolax® within 72 hours before the first dose of study drug.
21. Patient reports the use of rescue medication (Dulcolax®). for ≥3 days in either of the two weeks in the Pre-Treatment Assessment period.
22. Use of concomitant medications not allowed by the protocol prior to randomization。
23. Hospitalization for psychiatric disorder or suicide attempt within 2 years before the screening visit。
24. Patient reports participation in a clinical study within 30 days of the Screening visit or Five half-lives prior to visit 1.
25. Other circumstances in which the investigator considers the subject inappropriate for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Number of Durable Overall CSBM Responders, Mean Replacement Approach | 12-Week Treatment Period
  The primary efficacy endpoint will be the proportion of patients who are overall Complete spontaneous bowel movement (CSBM) responders during the 12-week Treatment Period. A CSBM weekly responder is defined as a patient who has ≥ 3 CSBMs per week and an increase from baseline of ≥ 1 CSBM for that week. An overall CSBM responder is a patient who is a weekly CSBM responder for at least 9 of the 12 treatment weeks, including at least 3 of the last 4 weeks.

SECONDARY OUTCOMES:
Change From Baseline in CSBMs (CSBMs/Week) Over the 12-week Treatment Period , Mean Replacement Approach | Baseline and 12 weeks
  The change from baseline in the number of Complete Spontaneous Bowel Movements (CSBMs) over the 12-week Treatment Period was analyzed. Baseline was the mean number of CSBMs recorded during the 2-week baseline diary assessment period prior to the first dose of study drug. A CSBM was a bowel movement that occurred in the absence of laxative use within 24 hours and was associated with the feeling of complete evacuation.
Change From Baseline in SBMs (SBMs/Week) Over the 12-week Treatment Period, Mean Replacement Approach | Baseline and 12 weeks
  The change from baseline in the number of Spontaneous Bowel Movement (SBM) over the 12-week Treatment Period was analyzed. Baseline was the mean number of SBMs recorded during the 2-week baseline diary assessment period prior to the first dose of study drug. The weekly SBM totals were derived from the daily diary entries reported during the Treatment Period.
Change From Baseline in Average Weekly SBM Stool Consistency Over the 12-week Treatment Period, Mean Replacement Approach | Baseline and 12 weeks
  The change from baseline in the stool consistency score (i.e. BSFS) over the 12-week Treatment Period was analyzed. Baseline was the mean BSFS score recorded during the 2-week baseline diary assessment period prior to the first dose of study drug. The weekly mean BSFS score per patient was derived from the BSFS entries reported during the Treatment Period in the Daily Symptom Diary.
  The stool consistency of each bowel movement (BM) was assessed by patients using the 7-point Bristol Stool Form Scale [BSFS] from 1 to 7.
  1. separate hard lumps like nuts (difficult to pass)
  2. sausage shaped but lumpy
  3. like a sausage but with cracks on its surface
  4. like a sausage or snake, smooth and soft
  5. soft blobs with clear-cut edges (passed easily)
  6. fluffy pieces with ragged edges, a mushy stool
  7. watery, no solid pieces (entirely liquid)
Change From Baseline in Average Weekly Straining Score Over the 12-week Treatment Period, Mean Replacement Approach | Baseline and 12 weeks
  The change from baseline in the straining score over the 12-week Treatment Period was analyzed. Baseline was the mean of non-missing straining scores recorded during the 2-week baseline diary assessment period prior to the first dose of study drug. The weekly average straining score was derived from the straining scores reported during the Treatment Period in the Daily Symptom Diary. The severity of straining during bowel movements was assessed on a 5-point Likert scale where 0 = none, 1 = mild, 2 = moderate, 3 = severe, and 4 = very severe.
Treatment Satisfaction | Baseline and 12 weeks
  For weeks 4, 8, and 12 (EOT), the treatment satisfaction question on Patient Global Assessment(PAG) questionnaires will be analyzed separately at each visit using an ANCOVA with fixed effects for gender (stratification variable) and treatment. (Grade 1-5; 1=none, 2=mild, 3=moderate, 4=severe, 5=very severe)
Time to First CSBMs and SBMs, Mean Replacement Approach | Baseline and 12 weeks
  Times to first CSBM and first SBM will be defined as the time from the first dose of study drug to the time of the first SBM and CSBM, respectively. Patients who have not had an SBM will be censored at the time of their first ingestion of rescue medication (not less than 72 hours after first dose of study drug) or at the time of Early Withdrawal, whichever is earlier.
  The primary analysis of time to first SBM will be to compare each plecanatide treatment versus placebo via a 2-sided log-rank test, stratified by gender. The functions of time to first SBM for each treatment group will be estimated using the K-M product-limit method. Two-sided, 95% CIs for median time to first SBM and other quartiles will be computed, by treatment group.
  A similar analysis will be done for time to first CSBM
Percent of Patients with an SBM within 24 Hours of the First Dose | Baseline and 12 weeks
  The percentage of patients with a SBM ≤24 hours after first dose will be analyzed using a Cochran-Mantel-Haenszel(test) (CMH) test stratified by gender to test the difference between each plecanatide group and placebo.
Percent of Patients with a CSBM within 24 Hours of the First Dose | Baseline and 12 weeks
  The percentage of patients with a CSBM ≤24 hours after first dose will be analyzed using a Cochran-Mantel-Haenszel(test) CMH test stratified by gender to test the difference between each plecanatide group and placebo.
Patient Reported Symptoms Associated With Constipation | Baseline and 12 weeks
  Patient-reported daily symptoms associated with constipation, measured using the 5-point score (0-4 rating), for the Treatment Period will be the average of non-missing patient scores by week, reported during that period. Comparisons will be made of changes from baseline for each parameter between each plecanatide treatment group and placebo, using a linear mixed-effect model under the assumption of normally distributed residuals with treatment group, week, interaction of treatment and week, gender and the corresponding baseline value as fixed effects and random intercept for patient.
Use of Rescue Medication | Baseline and 12 weeks
  Time to use of rescue medication will be defined as the time from the first dose of study drug to the time of the first use of provided rescue medication (Dulcolax®). Patients who haven't taken Dulcolax® will be censored at the time of their last rescue medication assessment or at the time of their Early Withdrawal, whichever is earliest.
Patient Global Assessments | Baseline and 12 weeks
  Patient Global Assessments include constipation severity, change in constipation symptoms and treatment assessments will be reported at (where applicable) Day 1 Pre-dose, Weeks, 4, 8, and 12 or (End of treatment) EOT and (End of study) EOS. Data will be summarized using descriptive statistics on observed data and change from baseline (where applicable). In addition, each assessment will be analyzed separately at each visit using an ANCOVA with fixed effects for gender (stratification variable) and treatment.
  In addition, a responder analyses based on change in constipation symptoms will be performed:
  Patient's response is minimally improved or better (i.e., score ≤ 3), or Patient's response is much improved or better (i.e., score ≤ 2)
Patient Assessment of Constipation- Quality of Life- (PAC-QOL©) | Baseline and 12 weeks
  Patient's QOL, measured using the 28-item PAC-QOL© questionnaires will be reported at Weeks 4, 8, and 12/EOT, and at the end of the Post-Treatment Period. Comparisons will be made of changes from baseline for the overall average of the 28 items between each plecanatide treatment and placebo using an ANCOVA model with treatment group and gender as fixed-effect terms, and the corresponding baseline value of the parameter as a covariate.
  The subscale scores (i.e., physical discomfort, psychosocial discomfort, worries/concerns, and satisfaction) will also be analyzed separately. For the measurements reported at the end of the Post-Treatment Period, additional comparisons will be made of changes from Week 12/EOT.
Patient Assessment of Constipation - Symptoms - (PAC-SYM©) | Baseline and 12 weeks
  Patient's symptoms, measured using the 12-item Patient Assessment of Constipation Symptoms（PAC-SYM© ）questionnaires will be reported at Weeks 4, 8, and 12 (EOT), and at the end of the Post-Treatment Period. Comparisons will be made of changes from baseline for the overall average of the 12 items between each plecanatide treatment and placebo using an ANCOVA model with treatment group and gender as fixed-effect terms, and the corresponding baseline value of the parameter as a covariate.
  The individual scores (e.g., discomfort in abdomen, pain in abdomen, etc.) will be also analyzed separately. For the measurements reported at the end of Post-Treatment Period, additional comparisons will be made of changes from Week 12/EOT.

OTHER OUTCOMES:
Safety Endpoints | Baseline and 12 weeks
  Evaluation of the safety of once daily plecanatide over 12 weeks of dosing will be based on the occurrence of Treatment emergent adverse event (TEAEs), vital signs, clinical laboratory assessments and, ECGs, and as compared with those noted in the placebo group.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No